CLINICAL TRIAL: NCT03770299
Title: A Phase 2 Multi-Center Randomized Trial to Assess Early Intervention With Adjuvant Nivolumab in Non-Small Cell Lung Cancer Participants With ctDNA-detected Minimal Residual Disease After Surgical Resection
Brief Title: An Investigational Immuno-therapy Study of Nivolumab Given After Surgery in Non-Small Cell Lung Cancer (NSCLC) Participants With Minimal Residual Disease
Acronym: CheckMate 9TN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9TN; 2018-003719-23 (EudraCT Number)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Circulating Tumor DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Vinorelbine; Gemcitabine; Docetaxel; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Nivolumab + SOC (chemotherapy in eligible participants or observation)
  Interventions: Biological: Nivolumab; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Docetaxel; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Other: Observation
- Arm B (Active Comparator): SOC (chemotherapy in eligible participants or observation)
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine; Drug: Docetaxel; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Other: Observation

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Arms: Arm A
Drug: Vinorelbine — Specified dose on specified days
Drug: Gemcitabine — Specified dose on specified days
Drug: Docetaxel — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days
Drug: Carboplatin — Specified dose on specified days
Drug: Paclitaxel — Specified dose on specified days
Other: Observation — Observation by the investigator

SUMMARY:
The purpose of this study is to determine if nivolumab added to the standard of care therapy (SOC) given after surgery is more effective than SOC alone in prolonging disease free survival in NSCLC participants with minimal residual disease detected after surgery.

ELIGIBILITY:
Inclusion Criteria prior to Surgery:

* Suspected or histologically confirmed Stage IIA to IIIB NSCLC with disease that is considered resectable
* Must be deemed eligible for complete resection and must agree to undergo standard of care surgery for complete resection of NSCLC
* Treatment naive (no previous systemic treatment)

Inclusion Criteria prior to Treatment Randomization:

* Must have undergone complete surgical resection of their Stage IIA to IIIB NSCLC
* Must have adequately recovered from surgery at the time of randomization
* Minimal residual disease (MRD) positive results as detected by ctDNA

Exclusion Criteria prior to Surgery:

* Participants with known EGFR mutations which are sensitive to available targeted inhibitor therapy (Prior to treatment randomization in select sites)
* Active, known or suspected autoimmune disease
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization

Exclusion Criteria prior to Treatment Randomization:

* Must continue to meet Exclusion Criteria prior to Surgery
* Must have no evidence of metastatic disease after surgery
* Received a live/attenuated vaccine within 30 days of first treatment

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2023-03-14 (Estimated); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Approximately 24 months

SECONDARY OUTCOMES:
Circulating tumor DNA (ctDNA) response rate | Approximately 36 months
ctDNA duration of response (DOR) | Approximately 36 months
ctDNA time to response (TTR) | Approximately 36 months
Incidence of adverse events (AEs) | Approximately 36 months
Incidence of serious adverse events (SAEs) | Approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm